CLINICAL TRIAL: NCT04968717
Title: 2000HIV Trained Innate Immunity in HIV Elite Controllers
Acronym: 2000HIVTrained
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Onze Lieve Vrouwe Gasthuis (Other); Elisabeth-TweeSteden Ziekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: NL76999.091.21; 2021-7495 (Other: Medical Ethics Committee CMO region Arnhem-Nijmegen)
Record Dates: First submitted 2021-04-13; First posted 2021-07-20 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Supernatants after PBMC stimulation experiments (no DNA) for assessment of cytokine production
  * Plasma for analysis of metabolomics and targeted proteomics (no DNA)
  * Cells for transcriptome analysis (contains DNA)
  * Cells prepared for epigenetic analyses (contains DNA)
  * DNA isolated for GWAS study (only in first-degree relative groups, contains DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV elite controllers: Non-viremic elite controller:
  HIV-positive , > 1 year without cART AND with >3 consecutive HIV-RNA < 75 copies/ml spanning >12 months AND stable CD4> 500 cells/uL.(i.e. >75% of measurements)
  OR on cART, but before start cART > 1 year without cART AND with >3 consecutive HIV-RNA < 75 copies/ml spanning >12 months AND stable CD4> 500 cells/uL. (i.e. >75% of measurements)
  Viremic elite controller:
  HIV-positive >5 year without cART AND with always HIV-RNA >50-10.000 copies/ml AND always CD4> 500 cells/uL.
  OR on cART, but before start cART >5 year without cART AND with always HIV-RNA >50-10.000 copies/ml AND always CD4> 500 cells/uL
- First-degree relatives of HIV elite controllers
- cART-treated non-controller HIV patients
- First-degree relatives of cART-treated non-controller HIV patients

SUMMARY:
Some individuals are able to spontaneously control HIV replication, the so-called 'elite controllers' (ECs). ECs are crucial for our understanding of HIV infection. While there is more and more evidence pointing towards a role of the innate immune system in elite control, no research has been performed on the role of innate trained immunity in elite control of HIV.

In this cross-sectional case-control study, we will study this role of trained immunity in HIV elite control by comparing ECs both to a non-HIV-infected first-degree relative, and to HIV patients who are not elite controllers. In addition, we will study whether HIV itself can induce a trained innate immunity phenotype.

DETAILED DESCRIPTION:
Rationale:

It remains unknown how some individuals spontaneously control HIV in the absence of antiretroviral medication, called HIV 'elite controllers' (ECs). ECs have been absolutely crucial to our current understanding of control of HIV replication. While research has mainly focused on the adaptive immune system, there is a vast amount of evidence indicating that the innate immune system is essential to HIV elite control.

Trained innate immunity can be expressed in terms of enhanced responsiveness of innate immune cells to a repeated trigger. This occurs through epigenetic remodeling after exposure to certain stimuli, such as beta-glucan, lipopolysaccharide (LPS) or the bacillus Calmette-Guérin (BCG) vaccine. Innate training results in an altered gene expression and metabolic reqiring on a cellular level, resulting in greater resistance against subsequent infection.

Both the impact of trained immunity on HIV infections and vice versa, the impact of HIV on trained immunity, are unknown. Our hypothesis is that ECs are natural hyper-responders to innate immune training triggers and that this aids in the HIV elite control phenotype.

Objectives:

1. (Primary) Investigate if a trained immunity profile in innate immune cells plays a role in HIV elite control.
2. (Secondary) Determine the immune phenotypes that distinguish family members of HIV elite controllers from family members of people living with HIV who have never been controllers.
3. (Secondary) Determine whether HIV can induce a long-term functional and transcriptional program in innate immune cells similar to trained immunity.

Study design:

Cross-sectional case-control study.

For the primary objective, HIV elite controllers will be compared to ART-suppressed HIV patients who never have been elite controllers and first-degree relatives of HIV elite controllers will be compared to first-degree relatives of ART-suppressed HIV patients who have never been elite controllers.

For the secondary objectives, first, a system biology approach will be used in the comparison above. To determine the role of HIV in trained innate immunity we will compare people living with HIV (both controllers as non-controllers) to their respective family members.

ELIGIBILITY:
All participants:

* All participants must be ≥18 years of age.
* Due to distorting effects on immune parameters and immune responses, participation is either not possible or must be delayed in case of the following:

  * active hepatitis B/C or signs of acute infections
  * active or recent malignant condition (i.e. <12 months ago treated)
  * active systemic auto-immune or auto-inflammatory conditions (such as rheumatoid arthritis, inflammatory bowel disease).
  * use of immunosuppressive medication
  * pregnant

HIV elite controllers:

HIV elite controllers in the 2000HIV that have an available first-degree relative. Definition of HIV elite controller is the same as in the 2000HIV, see definition on page 7 of the protocol and in the group description.

ART-suppressed people living with HIV:

As a control group, ART-suppressed people living with HIV in the 2000HIV that have an available first-degree relative will be included.

ART-suppressed people living with HIV need to apply to the following criteria to participate in the 2000HIV: ≥18 years, on cART ≥6 months with an HIV-RNA load <200 copies/mL.

For this 2000HIV-trained study, additional criteria for ART-suppressed people living with HIV are:

* Never applied to controller definition.
* At least one documented HIV RNA load >100.000 copies/mL
* No documentation of recent HIV acquisition combined with ART initiation in less than 6 months.

Eligible ART-suppressed people living with HIV will be matched by sex and age (max. 5-10 years apart), where possible. Similarity in family members between groups will also be pursued. That is why the HIV elite controllers and their family members will be enrolled first. Thereafter, the ART suppressed people living with HIV and their family members will be recruited and enrolled.

First-degree relatives:

Aside from the criteria for all participants mentioned above, there are no additional criteria for first-degree relatives of participants with HIV. If multiple first-degree relatives are available, siblings are preferred. If no sibling is available, then children >18 years. If no children >18 years, then parents. If there is still multiple options, same-sex will be preferred over different-sex relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A recent query of the Dutch national database of HIV (Athena Cohort; Stichting Hiv Monitoring (SHM)) revealed there are approximately 138 HIV elite controllers in the Netherlands, according to the definition used in the 2000HIV study. Of these, 80 HIV elite controllers are expected to participate in the 2000HIV study. Thanks to the query, each one of four 2000HIV participating centers is notified about who the HIV elite controllers in their center are. All HIV elite controllers participating in the 2000HIV will be approached and asked whether they have a first-degree relative who is available and willing to have a single venipuncture.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Direct cytokine responses | 24 hour ex vivo experiment
  Isolated monocytes and NK-cells will be stimulated ex vivo with a range of stimuli. Cytokines released in the supernatants will be measured by ELISA.
Cytokine responses after 6-day training | 7 day ex vivo experiment
  Isolated monocytes and NK-cells will be trained ex vivo and the innate training effect will be studied after restimulation with an unrelated stimulus on day 7. Cytokines released in the supernatant and intracellularly will be measured by ELISA.
Transcriptome | 1 year after sample collection
  RNA in the cells will be analysed to gain a transcriptional signature.
Epigenome | 1 year after sample collection
  Epigenetic signatures will be studied by means of ChIP sequencing and ATAC sequencing.
Immune phenotyping | 1 year after sample collection
  Circulating cells are phenotyped by menas of elaborate flow cytometry panels.

OTHER OUTCOMES:
Vaccination history | Collected during visit
  All groups
History of contracting COVID19 | Collected during visit
  All groups
Age | Collected during visit
  Only in first-degree relatives. Information on HIV patients already available from 2000HIV study (NCTNCT03994835).
Biological sex | Collected during visit
  Only in first-degree relatives. Information on HIV patients already available from 2000HIV study (NCTNCT03994835).
Medical history | Collected during visit
  Only in first-degree relatives. Information on HIV patients already available from 2000HIV study (NCTNCT03994835).
Medication use | Collected during visit
  Only in first-degree relatives. Information on HIV patients already available from 2000HIV study (NCTNCT03994835).

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - OLVG, Amsterdam
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided